CLINICAL TRIAL: NCT01228695
Title: Prospective Study of the Impact of Systemic Corticosteroid Use on Measures of Sleep Disordered Breathing
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israeli association for lung disease (Unknown)
Responsible Party: Israeli association for lung disease
Other Study IDs: IRB2421CTIL
Record Dates: First submitted 2010-10-21; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-02

CONDITIONS: Sleep Apnea
Keywords: steroids; patients treated with systemic steroids
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- steroid treatment
  Interventions: Other: sleep study

INTERVENTIONS:
Other: sleep study — The polysomnography (PSG) (Alice 3 System; Healthdyne, Atlanta, GA) consisted of continuous polygraphic recording from surface leads for electroencephalography, electrooculography, electromyography, electrocardiography, thermistors for nasal and oral airflow, thoracic and abdominal impedance belts for respiratory effort, pulse oximeter for oxyhemoglobin level, tracheal microphone for snoring, and sensors for leg and sleep position
  Other Names: no other names

SUMMARY:
Weight gain is both a significant risk factor for obstructive sleep apnea and a side-effect of long-term systemic steroids therapy.

This study aimed to investigate the impact of long-term systemic steroid treatment on sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, a scheduled therapy with a minimum daily dose of 10 mg prednisone (or equivalent) for at least 3 months was required

Exclusion Criteria:

* Patients younger than 18 years and those with known sleep apnea or other forms of sleep-disordered breathing were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for long-term treatment with oral prednisone (> 10 mg/d for 3 months or more)
Sampling Method: Non-Probability Sample
Enrollment: 20
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 3 months

SECONDARY OUTCOMES:
sleep study variables | 3 months
  apnea-hypopnea interval desaturation at the end of apnea interval snoring intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam health care campus, Haifa, Israel

REFERENCES:
- [Background] Yigla M, Tov N, Solomonov A, Rubin AH, Harlev D. Difficult-to-control asthma and obstructive sleep apnea. J Asthma. 2003 Dec;40(8):865-71. doi: 10.1081/jas-120023577. PMID 14736085